CLINICAL TRIAL: NCT01580306
Title: Pharmacokinetics, Safety and Tolerability of BI 201335 in Patients With Different Degrees of Renal Impairment in Comparison to Subjects With Normal Renal Function in a Monocentric, Open-label, Parallel-group, Phase I Trial
Brief Title: Pharmacokinetics and Safety of BI 201335 in Patients With Mild to Severe Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1220.58; 2011-005442-35 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-04-12; First posted 2012-04-19 (Estimated); Results first posted 2015-07-31 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — faldaprevir

ARMS (2):
- BI 201335 relevant treatment dose (A) (Experimental): Capsule for oral administration
  Interventions: Drug: BI 201335
- BI 201335 relevant treatment dose (B) (Experimental): Capsule for oral administration
  Interventions: Drug: BI 201335

INTERVENTIONS:
Drug: BI 201335 — Relevant treatment dose capsule (A) for oral administration
  Arms: BI 201335 relevant treatment dose (A)
Drug: BI 201335 — Relevant treatment dose capsule (B) for oral administration
  Arms: BI 201335 relevant treatment dose (B)

SUMMARY:
The main objective of this study is to investigate the influence of mild, moderate and severe renal impairment on the pharmacokinetics and safety of BI 201335 in comparison to a control group with normal renal function after single dose of BI 201335.

ELIGIBILITY:
Inclusion criteria:

Male and female healthy subjects with normal renal function and subjects with impaired renal function in relatively good health

Exclusion criteria:

Any relevant deviation from healthy conditions for healthy volunteers or significant diseases other than renal impairment for the renal impaired subjects

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1220.58.1 Boehringer Ingelheim Investigational Site, Kiel, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Renal Function: Capsule for oral administration (120 mg Faldaprevir)
  subjects with estimated glomerular filtration rate >= 90 mL/min/1.73m2
- Mild Renal Impairment: Capsule for oral administration (120 mg Faldaprevir)
  subjects with estimated glomerular filtration rate 60-89 mL/min/1.73m2
- Moderate Renal Impairment: Capsule for oral administration (120 mg Faldaprevir)
  subjects with estimated glomerular filtration rate 30-59 mL/min/1.73m2
- Severe Renal Impairment: Capsule for oral administration (120 mg Faldaprevir)
  subjects with estimated glomerular filtration rate 15-29 mL/min/1.73m2
Period: Overall Study
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Started | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (2.1) | 58.8 (9.3) | 67.1 (7.5) | 57.6 (9.5) | 61.4 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 3 | 11
  Male | 6 | 5 | 5 | 5 | 21

OUTCOME MEASURES:

1. Primary Outcome: AUC0-∞
Description: area under the concentration time curve of Faldaprevir in plasma over the time interval from 0 to infinity.
  In this endpoint, the data of AUC0-∞ show inter-individual variabilities.
Time Frame: 0:00, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 12:00,16:00, 24:00, 36:00, 48:00, 72:00, 96:00, 120:00, 144:00 hours (h) after administration
Population: Pharmacokinetic (PK) set: This subject set included all subjects in the treated set who provided at least 1 observation for at least 1 primary PK endpoint without important protocol violations relevant to the evaluation of PK, and who did not vomit at or before 2 times median tmax of unmetabolised faldaprevir.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 5 | 4 | 7 | 8
ng*h/mL | 76500 (95.7) | 86900 (89.8) | 136000 (67.2) | 129000 (98.8)
Statistical Analysis 1: Comparison: Normal Renal Function vs Mild Renal Impairment; relative bioavailability comparison mild : normal; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 113.57, 90% CI 2-sided [41.58 to 310.17], Standard Deviation 93.2 — the standard deviation is actually the geometric coefficient of variation
Statistical Analysis 2: Comparison: Normal Renal Function vs Moderate Renal Impairment; relative bioavailability comparison moderate : normal; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 178.31, 90% CI 2-sided [85.23 to 373.03], Standard Deviation 78.9 — the standard deviation is actually the geometric coefficient of variation
Statistical Analysis 3: Comparison: Normal Renal Function vs Severe Renal Impairment; relative bioavailability comparison severe : normal; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 169.21, 90% CI 2-sided [73.19 to 391.17], Standard Deviation 97.7 — the standard deviation is actually the geometric coefficient of variation

2. Primary Outcome: Cmax
Description: maximum concentration of Faldaprevir in plasma. In this endpoint, the data of Cmax show inter-individual variabilities.
Time Frame: 0:00, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 12:00,16:00, 24:00, 36:00, 48:00, 72:00, 96:00, 120:00, 144:00h after administration
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 5 | 4 | 7 | 8
ng/mL | 3810 (80.7) | 4080 (144.0) | 6680 (63.2) | 4600 (135.0)
Statistical Analysis 1: Comparison: Normal Renal Function vs Mild Renal Impairment; relative bioavailability comparison mild : normal; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 107.22, 90% CI 2-sided [35.16 to 327.01], Standard Deviation 107.7 — the standard deviation is actually the geometric coefficient of variation
Statistical Analysis 2: Comparison: Normal Renal Function vs Moderate Renal Impairment; relative bioavailability comparison moderate : normal; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 175.52, 90% CI 2-sided [89.55 to 344.06], Standard Deviation 70.4 — the standard deviation is actually the geometric coefficient of variation
Statistical Analysis 3: Comparison: Normal Renal Function vs Severe Renal Impairment; relative bioavailability comparison severe : normal; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 120.98, 90% CI 2-sided [47.257 to 309.736], Standard Deviation 115 — the standard deviation is actually the geometric coefficient of variation

3. Secondary Outcome: Clinical Relevant Abnormalities for Vital Signs, Physical Examination, Blood Chemistry, Haematology, Urinanalysis and ECG
Description: Clinical relevant abnormalities for Vital Signs, Physical Examination, Blood Chemistry, Haematology, Urinanalysis and ECG. New abnormal findings or worsening of baseline conditions were reported as Adverse Events.
Time Frame: from drug administration up to 2 weeks
Population: treated set
Measure: Number; unit: participants
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 8
participants
  Blood bilirubin increased | 0 | 0 | 0 | 1
  blood pressure systolic increased | 0 | 0 | 1 | 0

4. Secondary Outcome: Number of Participants With Drug Related Adverse Events
Description: number of participants with investigator-defined drug related adverse events.
Time Frame: drug administration until end-of-study examination (7 to 14 days after drug administration)
Population: treated set
Measure: Number; unit: participants
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 8
participants | 5 | 8 | 5 | 7

ADVERSE EVENTS:
Time Frame: From the time the subject signed the informed consent (21 days before drug administration) through the observational phase to the end of study visit (7 to 14 days after dosing)
Description: Subjects were required to report spontaneously any adverse events (AEs) as well as the time of onset, duration and intensity of these events. In addition, each volunteer was assessed regularly by the medical staff throughout the clinical trial as well as at the end of observation and whenever necessary as deemed by the investigator.
Groups:
- BI 201335 Relevant Treatment Dose (Normal Renal Function): Capsule for oral administration
  estimated glomerular filtration rate >= 90 mL/min/1.73m2
- BI 201335 Relevant Treatment Dose (Mild Renal Impairment): Capsule for oral administration
  estimated glomerular filtration rate 60-89 mL/min/1.73m2
- BI 201335 Relevant Treatment Dose (Moderate Renal Impairment): Capsule for oral administration
  estimated glomerular filtration rate 30-59 mL/min/1.73m2
- BI 201335 Relevant Treatment Dose (Severe Renal Impairment): Capsule for oral administration
  estimated glomerular filtration rate 15-29 mL/min/1.73m2
Arm/Group | BI 201335 Relevant Treatment Dose (Normal Renal Function) | BI 201335 Relevant Treatment Dose (Mild Renal Impairment) | BI 201335 Relevant Treatment Dose (Moderate Renal Impairment) | BI 201335 Relevant Treatment Dose (Severe Renal Impairment)
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 5/8 | 8/8 | 5/8 | 7/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 201335 Relevant Treatment Dose (Normal Renal Function) (N=8) | BI 201335 Relevant Treatment Dose (Mild Renal Impairment) (N=8) | BI 201335 Relevant Treatment Dose (Moderate Renal Impairment) (N=8) | BI 201335 Relevant Treatment Dose (Severe Renal Impairment) (N=8)
Diarrhoea (Gastrointestinal disorders) | 3 | 6 | 5 | 7
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 1 | 2
Vomiting (Gastrointestinal disorders) | 3 | 4 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1
Blood pressure systolic increased (Investigations) | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.